Desoximetasone Spray, 0.15%

Protocol / Study No. DSXS 1505 / 71542603

### STATISTICAL ANALYSIS PLAN

A Randomized, Double-Blind, Placebo-Controlled, Parallel-Design, Multiple-Site Clinical Study to Evaluate the Efficacy and Safety of Desoximetasone Topical Spray, 0.15% (Taro Pharmaceuticals, U.S.A., Inc.) in Patients with Mild to Moderate Plaque Psoriasis

Protocol Number: DSXS 1505 Novum Study Number: 71542603

### Sponsor:

Taro Pharmaceuticals U.S.A., Inc. 3 Skyline Drive, Hawthorne, NY 10532 USA

### **Contract Research Organization:**

Novum Pharmaceutical Research Services 225 W. Station Square Drive, Suite 200 Pittsburgh, PA 15219

March 4, 2016

Final Version 1.0

Desoximetasone Spray, 0.15%

Protocol / Study No. DSXS 1505 / 71542603

### **SAP Final Version Approvals**

A Randomized, Double-Blind, Placebo-Controlled, Parallel-Design, Multiple-Site Clinical Study to Evaluate the Efficacy and Safety of Desoximetasone Topical Spray, 0.15% (Taro Pharmaceuticals, U.S.A., Inc.) in Patients with Mild to Moderate Plaque Psoriasis

| Written By: Signature: Jianhua Liu, MSc Senior Biostatistician Novum Pharmaceutical Research Services | Date: 03/15/2016 |
|---|---|
| Reviewed By: Signature: Pina D'Angelo, MSc Senior Director, Scientific Affairs (Biostatistics) Novum Pharmaceutical Research Services | Date: 03/17/2016 |
| Approved By: Signature: Natalie Yantovskiy Director, Clinical Research Taro Pharmaceuticals U.S.A., Inc. | Date: 15 Man 2016 |

Desoximetasone Spray, 0.15% Protocol / Study No. DSXS 1505 / 71542603

### **Revision History**

| Version | DATE | DESCRIPTION OF REVISIONS | REVISED BY |
|-----------|-------------------|--------------------------|-------------|
| Draft 1.0 | February 18, 2016 | New Document | Jianhua Liu |
| Final 1.0 | March 4, 2016 | SAP Finalization | Jianhua Liu |

### Desoximetasone Spray, 0.15%

Protocol / Study No. DSXS 1505 / 71542603

### List of Abbreviations and Definition of Terms

ADaM Analysis Data Model

AE Adverse Event

ANCOVA Analysis of Covariance

BP Blood Pressure
BSA Body Surface Area

C Celsius

CRF Case Report Form

CDISC Clinical Data Interchange Standards Consortium

CRO Contract Research Organization

F Fahrenheit

FDA Food and Drug Administration

HR Heart Rate
Hg Mercury

ICF Informed Consent Form

ICH International Conference on Harmonization

IGA Investigator's Global Assessment

IND Investigational New Drug

LOCF Last Observation Carried Forward

MedDRA Medical Dictionary for Regulatory Activities

ITT Intent-to-Treat

LOCF Last Observation Carried Forward OGD The Office of Generic Drugs PASI Psoriasis Area Severity Index

PP Per-Protocol

SAE Serious Adverse Event
SAP Statistical Analysis Plan
SAS Statistical Analysis System
SDTM Study Data Tabulation Model
TLSS Total Lesion Severity Score
USA United States of America

### Desoximetasone Spray, 0.15% Protocol / Study No. DSXS 1505 / 71542603

### TABLE OF CONTENTS

| 1. | INTRODUCTION | 8 |
|---|---|---|
| 2. | OBJECTIVES | 8 |
| 3. | OVERALL STUDY DESIGN | 8 |
| 4. | RANDOMIZATION AND BLINDING | 12 |
| 5. | SAMPLE SIZE | 12 |
| | STUDY ENDPOINTS | |
| 7. | STUDY POPULATIONS | 14 |
| | STATISTICAL ANALYSIS METHODS | |
| | 8.1 Baseline Characteristics | 15 |
| | 8.1.1 Patient Disposition | 15 |
| | 8.1.2 Demographic and Other Baseline Characteristics | 15 |
| | 8.1.3 Medical History | |
| | 8.1.4 Concomitant Medications | |
| | 8.1.5 Pregnancy Test | 16 |
| | 8.2 Efficacy Analyses | |
| | 8.2.1 Primary Efficacy Analysis | |
| | 8.2.2 Secondary Efficacy Analysis | 16 |
| | 8.2.3 Treatment-by-Site Interaction and Pooling of Clinical Sites | 17 |
| | 8.3 Safety Analysis | 17 |
| | 8.3.1 Adverse Events | 17 |
| | 8.3.2 Vital Signs | 18 |
| | 8.3.3 Application Site Reactions | 18 |
| | 8.4 Multiple Comparisons | 18 |
| | 8.5 Methods for Handling Missing Data | 18 |
| | 8.6 Interim Analyses | 18 |
| 9. | TABLE, LISTING AND FIGURE SHELLS | 19 |
| | T16.1.9.1 Summary of Discontinued Patients | 21 |
| | T16.1.9.2 Summary of Protocol Deviations | 22 |
| | T16.1.9.3.1 Summary of Patients Excluded from Efficacy Analysis (Population | |
| | Determination) | 23 |
| | T16.1.9.3.2 Summary of Patients Included in Analysis Population by Study Center | 24 |
| | T16.1.9.4.1 Summary of Demographic Data | 25 |
| | T16.1.9.4.2 Summary of Baseline Dermatological Assessment | 2 <i>6</i> |
| | T16.1.9.5.1 Summary of Demographic Data (Intent-to-Treat Population) | 29 |
| | T16.1.9.5.2 Summary of Baseline Dermatological Assessment (Intent-to-Treat | |
| | Population) | |
| | T16.1.9.6.1 Summary of Demographic Data (Per-Protocol Population) | 29 |
| | T16.1.9.6.2 Summary of Baseline Dermatological Assessment (Per-Protocol | |
| | Population) | 29 |
| | T16.1.9.7.1 Summary of Frequency of Investigator Global Assessment (IGA) | 30 |
| | T16.1.9.7.2 Summary of Frequency of Investigator Global Assessment (IGA) | 31 |

| Desoximetasone Spray, 0.15% | Protocol / Study No. DSXS 1505 / 71542603 |
|-----------------------------|-------------------------------------------|

| TIC 1 0 0 1 C | |
|---|---|
| T16.1.9.8.1 Summary of Superiority Analysis Results of Co-Primary Efficacy | |
| Endpoint (Proportion of Patients in each Treatment that Have Clinical Success | 32 |
| ) ( | 52 |
| T16.1.9.8.2 Sensitivity Testing: Summary of Superiority Analysis Results of Co- | |
| Primary Efficacy Endpoint (Proportion of Patients in each Treatment that Have | 22 |
| Clinical Success based on IGA at Day 28±2) (Per-Protocol Population) | 3∠<br>22 |
| T16.1.9.9.1 Summary of Frequency of Total Lesion Severity Score (TLSS) | 3 |
| T16.1.9.9.2 Summary of Frequency of Total Lesion Severity Score (TLSS) (Per- | 33 |
| Protocol Population) | 3 |
| T16.1.9.10.1 Summary of Superiority Analysis Results of Co-Primary Efficacy | |
| Endpoint (Proportion of Patients in each Treatment that Have Treatment Success | 34 |
| based on TLSS at Day 28±2) (Intent-to-Treat Population) | 34 |
| T16.1.9.10.2 Sensitivity Testing: Summary of Superiority Analysis Results of Co- | |
| Primary Efficacy Endpoint (Proportion of Patients in each Treatment that Have | 24 |
| Treatment Success based on TLSS at Day 28±2) (Per-Protocol Population) | 34<br>25 |
| T16.1.9.11 Summary of Percent BSA Affected by Visit | 33 |
| T16.1.9.12 Summary of ANCOVA Analysis Results of Secondary Efficacy Endpoint | |
| (Change from Baseline in %BSA Affected at Day $28 \pm 2$ ) (Intent-to-Treat | 26 |
| Population) | 0د<br>77 |
| T16.1.9.13 Overall Summary of Adverse Events | 3 / |
| T16.1.9.14 Summary of Frequency of All Adverse Events by Body System (Safety | 38 |
| Population) | 30 |
| T16.1.9.15 Summary of Frequency of All Adverse Events by Relationship (Safety | 20 |
| 1 opulation, minimum minimum management and management management management and management managem | 39 |
| T16.1.9.16 Summary of Frequency of All Adverse Events by Severity (Safety | 40 |
| Population) | 40<br>41 |
| T16.1.9.17 Summary of Frequency of Serious Adverse Events (Safety Population) | 41<br>42 |
| T16.1.9.18 Summary of Adverse Events by Treatment (Safety Population) | 42 |
| T16.1.9.19 Summary of Vital Signs | 43<br>45 |
| L16.2.1 Listing of Discontinued Patients | |
| L16.2.2 Listing of Protocol Deviations | |
| L16.2.3 Patients Excluded from the Per-Protocol Population | 4 / |
| L16.2.4.1 Listing of Demographic Data | 48 |
| L16.2.4.2 Listing of Medical History | 49 |
| L16.2.4.3 Listing of Concomitant Medication | |
| L16.2.5.1 Listing of Visit Date Information | |
| L16.2.5.2 Listing of Drug Administration | |
| L16.2.5.3 Listing of Study Medication Weight | |
| L16.2.6.1 Listing of Investigator Global Assessment (IGA) | 54 |
| L16.2.6.2 Listing of Total Lesion Severity Score (TLSS) | 55 |
| L16.2.6.3 Listing of Psoriasis Area Severity Index (PASI), Target Lesion size and | |
| BSA Affected | 56 |
| L16.2.6.4 Listing of Investigator Evaluator Initials | 57 |

| Desoximetasone Spray, 0.15% | Protocol / Study No. DSXS 1505 / 715 | <u>42603</u> |
|---|---|---|
| L16.2.7.1 Listing of Adverse Events by | Freatment | 58 |
| · | action | |
| | ults | |
| • | | |
| Appendix A: Total Body Surface Area C | alculation | 62 |
| | (TLSS) | |
| | ssment (IGA) | |
| | ex (PASI) | |
| * * | | |

Desoximetasone Spray, 0.15%

Protocol / Study No. DSXS 1505 / 71542603

### 1. INTRODUCTION

This Statistical Analysis Plan (SAP) is based on the final Clinical Study Protocol DSXS 1505 (Novum Study No. 71542603) Rev. 4 dated 02/24/2016. The SAP provides details on the planned statistical methodology for the analysis of the study data. The SAP also outlines the statistical programming specifications for the tables, listings and figures.

This SAP describes the study endpoints, derived variables, anticipated data transformations and manipulations, and other details of the analyses not provided in the study protocol. This SAP therefore outlines in detail all other aspects pertaining to the planned analyses and presentations for this study.

The following documents were reviewed in preparation of this SAP:

- Final Clinical Study Protocol DSXS 1505 (Novum Study No. 71542603) Rev. 4 dated 02/24/2016
- Case Report Form Booklet Version 1.0 for Novum Study No. 71542603 dated September 3, 2015

The reader of this SAP is encouraged to also read the clinical protocol for details on the conduct of this study, and the operational aspects of clinical assessments and timing for completing a patient in this study.

### 2. OBJECTIVES

To evaluate the therapeutic efficacy and safety of desoximetasone topical spray, 0.15% (Taro Pharmaceuticals, U.S.A., Inc.) compared to a Placebo (vehicle) spray (Taro Pharmaceuticals, U.S.A., Inc.) in patients with mild to moderate plaque psoriasis.

### 3. OVERALL STUDY DESIGN

This double-blind, randomized, placebo-controlled, parallel group, multi-site study is designed to evaluate the therapeutic efficacy and safety of desoximetasone topical spray, 0.15% (Taro Pharmaceuticals, U.S.A., Inc.).

Up to 120 patients will be enrolled to randomize up to 60 patients in the Test group and 60 in the Placebo group. Before any study-specific procedures are performed all patients will read and sign the IRB-approved informed consent form. In addition, patients considered as minors by the state law in which the clinical site is located (in most States under 18 years of age), must have a signed parental/guardian Informed Consent Form (ICF), indicating approval to participate, as well as a signed assent to participate form.

### Desoximetasone Spray, 0.15%

Protocol / Study No. DSXS 1505 / 71542603

To qualify for inclusion in the study, patients must be at least 12 years of age with a confirmed diagnosis of mild to moderate plaque psoriasis and must fulfill the following primary inclusion criteria:

- An affected BSA of 5 10% (Appendix A)
- A IGA score of 2 (mild) or 3 (moderate) (Appendix B)
- Target Lesion area of at least 5 cm<sup>2</sup>
- Plaque Elevation Score ≥ 2 for the Target Lesion (based on TLSS score, Appendix B)

At Visit 1, patients who meet all inclusion/exclusion criteria will be randomized in a 1:1 ratio (Test: Placebo) for 28 days of treatment:

- Test: Desoximetasone topical spray, 0.15% (Taro Pharmaceuticals, U.S.A., Inc.)
- Placebo: Vehicle spray (Taro Pharmaceuticals, U.S.A., Inc.)

Randomized study medication will be self-administered by the patient for 28 days. Patients will be instructed to spray the study medication directly to all affected areas and gently and completely rub in the study drug twice a day for 28 days. Study medication will be applied in the morning and evening approximately 12 hours apart. Patients will return to the clinic at scheduled Visits 2, 3 and 4. Each patient will be provided with a dosing diary in which they will be required to record dosing dates and times. These diaries should be brought to each visit so that the study staff may check compliance. At the end of the study, the dosing diaries will be retained in the patient's file as source documentation.

During the study patients will visit the research center for a total of 4 scheduled visits:

- Visit 1: Randomization (Day 1),
- Visit 2: Interim Visit (Day  $7 \pm 2$ ),
- Visit 3: Interim Visit (Day  $14 \pm 2$ ),
- Visit 4: End of Treatment (Day  $28 \pm 2$ ).

Patients will be contacted at Day  $42 \pm 4$  (Visit 5) for a Telephone Follow-up to report any Adverse Events that have occurred since the end of treatment,

Evaluation of therapeutic efficacy will be primarily based on dermatological evaluation of psoriasis. The evaluation will include scoring of the extent and severity of plaque psoriasis. Refer to Appendices A, B and C for body surface area (BSA) estimation, Investigator's Global Assessment Scale (IGA), Total Lesion Severity Score (TLSS) and Psorasis Area Score Index

Desoximetasone Spray, 0.15% Protocol / Study No. DSXS 1505 / 71542603

(PASI), respectively. Selected sites will be instructed to take photographs of a target lesion at each visit.

Desoximetasone Spray, 0.15%

Protocol / Study No. DSXS 1505 / 71542603

**Figure 1 Study Schematic** 

| PROCEDURE | VISIT 1<br>Randomization<br>Day 1 | VISIT 2<br>Interim<br>Visit<br>Day 7<br>± 2 days | VISIT 3 Interim Visit Day 14 ± 2 days | VISIT 4 End of Treatment Day 28 ± 2 days | VISIT 5 Telephone Follow-Up Visit Day 42 ± 4 days |
|---|---|---|---|---|---|
| Informed Consent | X | | | | |
| Medical History & Demographics | X | | | | |
| Height and Weight | X | | | | |
| Vital Signs | X | X | X | X | |
| Dermatological<br>Assessment | X | X | X | X | |
| % BSA Assessment | X | X | X | X | |
| IGA Score | X | X | X | X | |
| Total Lesion<br>Severity Score | X | X | X | X | |
| PASI Score | X | X | X | X | |
| Application Site<br>Reactions | X | Х | X | X | |
| Target Lesion Photograph** | Х | X | X | X | |
| Pregnancy Test* | X | | | X | |
| Concomitant<br>Medication | X | X | X | X | |
| Collect/Dispense<br>Study Medication | X | | X | X | |
| Provide/Review patient Dosing Diary | Х | X | X | Х | |
| Adverse Events | | X | X | X | X |
| Evaluation of Patient Compliance to the Protocol | | Х | X | Х | |

<sup>\*</sup> Pregnancy Test will be conducted for women of child-bearing potential

\*\* Selected sites will be designated to take photographs of a defined target lesion at each Clinic Visit

Desoximetasone Spray, 0.15%

Protocol / Study No. DSXS 1505 / 71542603

### 4. RANDOMIZATION AND BLINDING

The study drug will be randomized, packaged and blinded by an independent packaging company. Randomization will be pre-planned according to a computer-generated randomization schedule. The randomization will be generated in blocks, each containing 4 patients' worth of medication (2 x Test product and 2 x Placebo). Each patient kit will contain 2 x 100 ml bottles of study medication.

The randomization number will be a unique 4 digit number.

A perforated or two-part label will be attached to the box of drug supplies for each patient. Both pieces of the label should include the following information: protocol number, randomization number, space for patient's initials, statement that the drug is for Investigational Use Only, space for dispensing date, storage information and the Sponsor's name. One part of the label shall remain attached to the box. The other part will be removed before dispensing and attached to the patient's source documents.

At the end of the study, after all the clinical data have been entered and the study database has been locked, a copy of the randomization will be sent to the statistician.

The Investigator, staff at the study site, study monitors, and data analysis/management personnel will be blinded to the patient assignment.

### 5. SAMPLE SIZE

The primary analyses of interest are the proportion of patients in the Test and Vehicle treatment groups who are considered to be a Clinical Success and Treatment Success on Day 28.

In-house data from two Phase III studies that evaluated the safety and efficacy of desoximetasone spray 0.25% (twice daily for 28 days) in patients with moderate to severe plaque psoriasis were used for sample size determination. These studies were conducted in support of Taro's NDA #204141, Topicort® (desoximetasone) Topical Spray, 0.25%. In those studies the Clinical Success rates were 31% and 53% for the active product (42% average) and 5% and 18% for the vehicle treatment (12% average), and the Treatment Success rates were 39% and 53% for the active product (46% average) and 7% and 17% for the vehicle treatment (12% average).

Based on the average results from these two studies on the 0.25% spray, the proportion of subjects in the Test group considered a Clinical Success and Treatment Success is expected be 40% or higher and the proportion of subjects in the Vehicle group considered a Clinical Success and Treatment Success is expected to be 12% or less for desoximetasone spray 0.15% in patients with mild to moderate plaque psoriasis. With these assumptions, 50 evaluable subjects in the ITT in each treatment group will demonstrate superiority of the Test to the Vehicle group with 89% power

### Desoximetasone Spray, 0.15%

Protocol / Study No. DSXS 1505 / 71542603

at the 5% level of significance (p < 0.05, using two-sided Z-test), assuming 100% correlation between Clinical and Treatment Success rates.

To allow for patients who may drop out from the study or are otherwise non-evaluable, up to 120 patients may be enrolled (60 in the Test group and 60 in the Vehicle group).

### 6. STUDY ENDPOINTS

### **Primary Efficacy Endpoints**

- 1. The proportion of patients in each treatment group who are considered a Clinical Success at Day  $28 \pm 2$  (i.e., at least a 2-grade improvement from the patient's baseline IGA score)
- 2. The proportion of patients in each treatment group who are considered a Treatment Success for the Target Lesion at Day  $28 \pm 2$  (i.e., a TLSS value of 0 or 1 at Day  $28 \pm 2$  for each of the three signs and symptoms (i.e., erythema, scaling and plaque elevation) depending on the patient's baseline TLSS)

### **Definitions:**

- 1. <u>Treatment Success:</u> To be considered a Treatment Success the patient's TLSS value at Day  $28 \pm 2$  must be 0 if their baseline TLSS value is 2 and must be 0 or 1 if their baseline TLSS value is > 2 for each of the individual signs and symptoms
- 2. <u>Treatment Failure:</u> A patient will be considered a Treatment Failure if:
  - a. the patient's TLSS value is > 0 if their baseline TLSS value is 2 or > 1 if their baseline IGA score is > 2 for any of the individual signs and symptoms
  - b. the patient was considered to have an insufficient therapeutic response
- 3. <u>Clinical Success:</u> To be considered a Clinical Success the patient must have at least a 2-grade improvement from their baseline IGA score. That is, an IGA score of 0 at Day 28 ± 2 if their baseline IGA score is 2 or an IGA score of 0 or 1 at Day 28 ± 2 if their baseline IGA score is 3
- 4. Clinical Failure: A patient will be considered a Clinical Failure if:
  - a. the patient's IGA score is > 0 if the baseline IGA score is 2 or > 1 if the baseline IGA score is 3
  - b. the patient was considered to have an insufficient therapeutic response

### **Secondary Efficacy Endpoint**

The change from baseline in %BSA affected at Day  $28 \pm 2$ 

Desoximetasone Spray, 0.15%

Protocol / Study No. DSXS 1505 / 71542603

### 7. STUDY POPULATIONS

### Intent-to-Treat (ITT) Population

The ITT population will include:

• All randomized subjects.

Patients discontinued early for any reason will be included in the ITT with their Last Observation Carried Forward (LOCF).

### Per-Protocol (PP) Population

The PP population is a sub-population of the ITT population and will include:

- Patients who met all inclusion and exclusion criteria and were randomized according to the randomized treatment assignment.
- Patients who applied at least one dose AND had at least one post-baseline evaluation.
- Patients who were compliant with the dosage regimens following randomization.
- Patients who had no major protocol deviations.

### Safety Population

• All patients who were randomized and received at least one dose of the study product.

### 8. STATISTICAL ANALYSIS METHODS

If not otherwise specified, statistical significance is defined as p<0.05 and is two-tailed. Data will be summarized with respect to demographic and baseline characteristics and safety variables.

For categorical variables, the number and percent of each category within a parameter will be calculated for non-missing data. For continuous variables, statistics will include n, mean, standard deviation, median, minimum and maximum values.

All statistical analyses will be conducted using SAS<sup>®</sup>, Version 9.4 or higher. Datasets will be prepared using headings from Clinical Data Interchange Consortium (CDISC) Study Data Tabulation Model (SDTM) implementation for human clinical trials and ADaM (Analysis Dataset Model).

Desoximetasone Spray, 0.15%

Protocol / Study No. DSXS 1505 / 71542603

### 8.1 Baseline Characteristics

### 8.1.1 Patient Disposition

The patient disposition information will be summarized by treatment. The number of patients randomized, treated with study medication will be tabulated by treatment. In addition, completion status and primary reason for withdrawal will be summarized by treatment.

### 8.1.2 Demographic and Other Baseline Characteristics

Baseline comparability of all treatment groups will be evaluated separately in the ITT, PP and Safety populations.

The following baseline demographics (determined from their initial study visit) will be evaluated:

- Age (years)
- Gender (male/female)
- Ethnicity (Hispanic/non Hispanic)
- Race (White, Black/African American, Native Hawaiian or Other Pacific Islander, Asian, American Indian or Alaska Native, Other)
- Baseline total BSA
- Baseline % BSA affected with psoriasis
- IGA score
- TLSS Score
- PASI Score
- Target Lesion size (area)

Summary tables by treatment will be presented. Continuous variables will be summarized using descriptive statistics (n, mean, standard deviation, median, minimum, maximum). Categorical variables will be summarized using frequencies and percentage.

Baseline comparability of the treatments will be presented using Chi-square test for the categorical variables, and Analysis of Variance for the continuous variables.

All data will be listed by treatment and patient.

### 8.1.3 Medical History

At Visit 1 patients will be questioned about personal medical history including psoriasis history

### Desoximetasone Spray, 0.15%

Protocol / Study No. DSXS 1505 / 71542603

and all medication use within the previous 12 weeks.

Medical history data will be listed by treatment and patient.

### **8.1.4 Concomitant Medications**

At each clinic visit, patients will be questioned about current and concomitant medication use. Patients will also be questioned about ongoing or new concomitant medication use during the treatment period at Visits 2, 3 and 4.

All prior and concomitant medications taken since screening until the end of the study will be listed by treatment and patient.

### 8.1.5 Pregnancy Test

All females of childbearing potential will have a urine pregnancy test performed at Visit 1 and Visit 4.

Pregnancy test results will be listed by treatment and patient.

### 8.2 Efficacy Analyses

### 8.2.1 Primary Efficacy Analysis

The primary endpoints are: 1) the proportion of patients in each treatment group who are considered a Clinical Success at Day  $28 \pm 2$  (i.e., at least a 2-grade improvement from the patient's baseline IGA score). 2) the proportion of patients in each treatment group who are considered a Treatment Success for the Target Lesion at Day  $28 \pm 2$  (i.e., a TLSS value of 0 or 1 at Day  $28 \pm 2$  for each of the three signs and symptoms (i.e., erythema, scaling and plaque elevation) depending on the patient's baseline TLSS).

The Test treatment will be compared with Placebo for each primary endpoint at the 5% significance level (p < 0.05; using two-tailed Z-test) in the ITT population using last observation carried forward (LOCF). Superiority of Test over Placebo will be demonstrated if both dichotomous endpoints show statistical significance at the 5% significance level by the Z-tests.

For sensitivity testing, the primary analysis will also be performed using the PP population.

### 8.2.2 Secondary Efficacy Analysis

The secondary endpoint is the change from baseline in %BSA affected at Day  $28 \pm 2$ .

The Test treatment will be compared with Placebo for the secondary endpoint at the 5% significance level in the ITT population using LOCF. Analysis of Covariance (ANCOVA) with

### Desoximetasone Spray, 0.15%

Protocol / Study No. DSXS 1505 / 71542603

treatment and site as fixed effects and baseline %BSA as a covariate in the model will be used for the evaluation of the secondary endpoint.

The LSMeans for each treatment, the LSMeans of the treatment difference together with the corresponding 95%-confidence interval and the p-value will be presented.

Descriptive statistical analysis (number of patients, mean, standard deviation, median, minimum and maximum) will be generated to compare the efficacy results in each treatment group at each visit.

### 8.2.3 Treatment-by-Site Interaction and Pooling of Clinical Sites

As this is a multiple-site study, the interaction of treatment-by-site may be evaluated for superiority testing by the Cochran-Mantel-Haenszel test (stratified by site) for the primary efficacy endpoints and by ANCOVA for the secondary endpoint at the 5% significance level (p < 0.05, 2-sided) in the ITT population. A site(s) with a low enrollment rate(s) may be pooled with its geographically closest site, so as to avoid bias in the estimation of a treatment-by-site interaction effect. The pooling will be done for low enrolling sites that account for less than 4-7% of the total number of patients in the ITT population at the site with the highest enrolling rate. If no treatment-by-site interaction is identified with the primary endpoints then no adjustment will be made to any efficacy analysis and treatment-by site interaction will not be included as a term in the statistical models for evaluating superiority.

### 8.3 Safety Analysis

Safety analysis will be conducted on safety population.

### 8.3.1 Adverse Events

All the adverse events (AEs) reported throughout the study will be coded and classified according to the MedDRA (Medical Dictionary for Regulatory Activities) coding dictionary (Version 17.0 or higher). Each adverse event is to be evaluated for date of start and end, seriousness, severity, causal relationship with the study drugs, action taken and outcome.

All AEs will be listed by treatment and patient.

A summary table of the number and percent of patients with AEs by system organ class, preferred term, and treatment will be presented. Each patient will be counted only once within each preferred term.

A frequency summary table of the number of AEs by system organ class, preferred term, severity, and treatment will be presented. Severity will be classified as "Mild", "Moderate", or "Severe".

### Desoximetasone Spray, 0.15%

Protocol / Study No. DSXS 1505 / 71542603

Similarly, a frequency summary table of the number of AEs by system organ class, preferred term, and relationship to a study drug, and treatment will be presented. Relationship to a study drug will be classified as "Not Related" or "Related" where "Related includes "Possible", "Probable", or "Definite".

Should sufficient data exist, adverse event frequencies will be compared between treatments using Fisher's exact test.

### 8.3.2 Vital Signs

The patient's vital signs will be recorded (heart rate, blood pressure, temperature and respiration rate) at Visit 1, 2, 3 and 4.

Descriptive summaries (number of observations, mean, standard deviation, minimum, median and maximum) will be provided by treatment and visit.

All data will be listed by treatment and patient.

### 8.3.3 Application Site Reactions

At each visit the Investigator will examine the treatment area and complete the signs and symptoms of irritation assessment based on the scale provided in Appendix E.

A frequency summary table comparing the application site reactions for each treatment group will be presented by visit.

All data will be listed by treatment and patient.

### 8.4 Multiple Comparisons

No multiple comparison adjustment will be made in this study.

### 8.5 Methods for Handling Missing Data

For demographic and baseline characteristics, each variable will be analyzed using all available data. Patients with missing data will be excluded only from analyses for which data are not available.

For primary and secondary efficacy analysis, patients discontinued early for any reason will be included in the ITT with their Last Observation Carried Forward (LOCF).

### 8.6 Interim Analyses

There is no interim analysis planned in this study.

Desoximetasone Spray, 0.15%

Protocol / Study No. DSXS 1505 / 71542603

### 9. TABLE, LISTING AND FIGURE SHELLS

The following shells are provided in order to provide a framework for the display of data from this study. These shells may not be reflective of every aspect of this study but are intended to show the general layout of the Tables, Listings and Figures that will be included in the final clinical study report. Tables, Listings and Figures are numbered following the ICH structure. Table headers, variables names and footnotes will be modified as needed following data analyses. All descriptive and inferential statistical analyses will be performed using SAS® statistical software Version 9.4 or higher, unless otherwise noted.

TABLE, LISTING AND FIGURE SHELLS

■ Taro Pharmaceuticals U.S.A., Inc ■

T16.1.9.1 Summary of Discontinued Patients

Taro Pharmaceuticals U.S.A., Inc

Desoximetasone Spray, 0.15%

Novum Pharmaceutical Research Services Protocol / Study No. DSXS 1505 / 71542603

| | | | XXX |
|---------------------------------------------------------|---|-----|-----|
| | Ų | XXX | XXX |
| | V | XXX | XXX |
| l erminated Early xxx | ~ | XXX | XXX |
| Early Termination Reason | ~ | XXX | XXX |
| Adverse Event xxx | ~ | XXX | XXX |
| Insufficient therapeutic response/treatment failure xxx | v | xxx | XXX |
| Lost to follow-up | ~ | XXX | XXX |
| etc. | | | |
| Other | × | XXX | XXX |

T16.1.9.2 Summary of Protocol Deviations

Taro Pharmaceuticals U.S.A., Inc Desoximetasone Spray, 0.15%

Novum Pharmaceutical Research Services Protocol / Study No. DSXS 1505 / 71542603

| | Test: Desoximetasone Topical spray, 0.15% | Placebo: Vehicle<br>spray | Total |
|---|---|---|---|
| Total Patients with Protocol Deviations | XXX | XXX | XXX |
| Total Deviations | XXX | XXX | XXX |
| Lost to Follow-up | XXX | XXX | XXX |
| Missed Visit | XXX | XXX | XXX |
| Missed more than 3 consecutive days of dosing | XXX | XXX | XXX |
| Non-compliance with dosing requirements | XXX | XXX | XXX |
| Outside Visit Window | XXX | XXX | XXX |
| Restricted Medication Use | XXX | XXX | XXX |
| Randomized in Error | XXX | XXX | XXX |
| Other | XXX | XXX | XXX |

Path: L:\Studies\_Sas\_Codes\Clinical Trial\71542603\PDF\xxx Created on: ddmmmyy hh:mm

T16.1.9.3.1 Summary of Patients Excluded from Efficacy Analysis

Taro Pharmaceuticals U.S.A., Inc Desoximetasone Spray, 0.15%

Novum Pharmaceutical Research Services Protocol / Study No. DSXS 1505 / 71542603

(Population Determination)

| | l'est: | Disease | |
|---|---|---|---|
| | Desoximetasone<br>Topical spray, 0.15% | Flacebo:<br>Vehicle spray | Total |
| Randomized / ITT Population | XXX | XXX | XXX |
| Safety Population | XXX | XXX | XXX |
| PP Population | XXX | XXX | xxx |
| Excluded from PP population | XXX | XXX | XXX |
| Inclusion/Exclusion criteria not met | XXX | XXX | XXX |
| Non-compliant with dosing requirement | XXX | XXX | XXX |
| Major protocol deviations | XXX | XXX | XXX |
| etc. | XXX | XXX | XXX |
| | XXX | XXX | xxx |

■ Taro Pharmaceuticals U.S.A., Inc ■

Novum Pharmaceutical Research Services Protocol / Study No. DSXS 1505 / 71542603 T16.1.9.3.2 Summary of Patients Included in Analysis Population by Study Center

| | | PPP | | | ITT | | | Safety | |
|---|---|---|---|---|---|---|---|---|---|
| Total<br>Randomized | Test | Placebo | Total | Test | Placebo | Total | Test | Placebo | Total |
| XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | xxx | XXX |
| XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |

Path: L:\Studies\_Sas\_Codes\Clinical Trial\71542603\PDF\xxx Created on: ddmmmyy hh:mm


T16.1.9.4.1 Summary of Demographic Data

Taro Pharmaceuticals U.S.A., Inc Desoximetasone Spray, 0.15%

Novum Pharmaceutical Research Services Protocol / Study No. DSXS 1505 / 71542603

| | | Test: Desoximetasone Topical spray, 0.15% N=xx | Placebo:<br>Vehicle spray<br>N=xx | Total<br>N=xx | P-value |
|---|---|---|---|---|---|
| Age (years) | u | XX | XX | XX | X.XXXX |
| | Mean ± SD | $XX.X \pm X.X$ | $XX.X \pm X.X$ | $XX.X \pm X.X$ | |
| | Median | XX.X | XXX.X | XX.X | |
| | Range | XX-XX | XX-XX | XX-XX | |
| Age Groups | < 18 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | X.XXXX |
| | 18 – 40 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| | 41 - 64 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| | 65 - 75 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| | > 75 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Race | American Indian or Alaska Native | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | X.XXXX |
| | Asian | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| | Black/African American | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| | Native Hawaiian or other Pacific<br>Islander | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| | White | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| | Other | $XX (XX.X^{9/6})$ | xx (xx.x%) | xx (xx.x%) | |
| Ethnicity | Hispanic or Latino | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | X.XXXX |
| | Not Hispanic or Latino | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Gender | Female | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | X.XXXX |
| | Male | XX (XX.X%) | xx (xx.x%) | xx (xx.x%) | |

N= number of patients in the treatment; n= number of patient with data available; % is based on N

Protocol / Study No. DSXS 1505 / 71542603

Taro Pharmaceuticals U.S.A., Inc Desoximetasone Spray, 0.15%

Novum Pharmaceutical Research Services

| Assessment |
|----------------|
| 7 |
| <u>ت</u> |
| 5 |
| 2 |
| atological |
| a |
| Ξ |
| Ξ |
| ě |
| ine |
| <u>-</u> |
| f Base |
| × |
| £B |
| 5 |
| > |
| = |
| 13 |
| Ξ |
| Ξ |
| Ξ |
| ij |
| 4 |
| Ò |
| T16.1.9.4.2 Su |
| 6 |
| T16 |

| | | Test: Desoximetasone Topical spray, 0.15% N=xx | Placebo:<br>Vehicle spray<br>N=xx | Total<br>N=xx | P-value |
|---|---|---|---|---|---|
| Baseline Total BSA | ч | XX | XX | XX | X.XXXX |
| | Mean ± SD | $XX.X \pm X.X$ | $XX.X \pm X.X$ | $xx.x \pm x.x$ | |
| | Median | XX.X | XX.X | XXX.X | |
| | Range | XX-XX | XX-XX | xx-xx | |
| % BSA Affected with Psoriasis | и | XX | XX | XX | X.XXXX |
| | Mean ± SD | $XX.X \pm X.X$ | $XX.X \pm X.X$ | $XX.X \pm X.X$ | |
| | Median | XX.X | XX.X | XX.X | |
| | Range | XX-XX | XX-XX | XX-XX | |
| Baseline IGA Score | Clear | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | X.XXXX |
| | Minimal | XX (XX.X%) | xx (xx.x%) | xx (xx.x%) | |
| | Mild | xx (xx.x%) | xx (xx.x%) | xx (xx.x <sup>9</sup> %) | |
| | Moderate | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| | Severe | (%X:XX) XX | xx (xx.x%) | xx (xx.x%) | |

N= number of patients in the treatment; n= number of patient with data available; % is based on N


T16.1.9.4.2 Summary of Baseline Dermatological Assessment

Novum Pharmaceutical Research Services Protocol / Study No. DSXS 1505 / 71542603

| | | l est: Desoximetasone Topical spray, 0.15% N=xx | Placebo:<br>Vehicle spray<br>N=xx | Total<br>N=xx | P-value |
|---|---|---|---|---|---|
| Baseline TLSS | Clear | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | X.XXXX |
| | Almost Clear | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| | Mild | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| | Moderate | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| | Severe | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| | Very Severe | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Baseline Scaling Score | Clear | XX (XX.X%) | xx (xx.x%) | xx (xx.x%) | X.XXXX |
| | Almost Clear | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| | Mild | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| | Moderate | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| | Severe | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| | Very Severe | XX (XX.X%) | xx (xx.x%) | xx (xx.x%) | |
| Baseline Erythema Score | Clear | XX (XX.X%) | xx (xx.x%) | xx (xx.x%) | X.XXXX |
| | Almost Clear | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| | Mild | XX (XX.X%) | xx (xx.x%) | xx (xx.x%) | |
| | Moderate | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| | Severe | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| | Very Severe | xx (xx.x%) | (%X:XX) XX | xx (xx.x%) | • |

N= number of patients in the treatment; n= number of patient with data available; % is based on N

Taro Pharmaceuticals U.S.A., Inc Desoximetasone Spray, 0.15%

T16.1.9.4.2 Summary of Baseline Dermatological Assessment

Novum Pharmaceutical Research Services Protocol / Study No. DSXS 1505 / 71542603

| | | Test: Desoximetasone Topical spray, 0.15% N=xx | Placebo:<br>Vehicle spray<br>N=xx | Total<br>N=xx | P-value |
|---|---|---|---|---|---|
| Baseline Plaque Elevation | Clear | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | X.XXXX |
| | Almost Clear | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| | Mild | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| | Moderate | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| | Severe | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| | Very Severe | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Baseline PASI Score | п | XX | XX | XX | X.XXXX |
| | $Mean \pm SD$ | $XX.X \pm X.X$ | $XX.X \pm X.X$ | $XX.X \pm X.X$ | |
| | Median | XX.X | XX.X | XX.X | |
| | Range | XX-XX | XX-XX | XX-XX | |
| Target Lesion Size (area, cm^2) | u | XX | XX | xx | X.XXX |
| | $Mean \pm SD$ | $XX.X \pm X.X$ | $XX.X \pm X.X$ | $XX.X \pm X.X$ | |
| | Median | XX.X | XX.X | XX.X | |
| | Range | XX-XX | XX-XX | xx-xx | |
| Baseline PASI Score | u | XX | XX | XX | X.XXXX |

N= number of patients in the treatment; n= number of patient with data available; % is based on N

Path: L:\Studies\_Sas\_Codes\Clinical Trial\71542603\PDF\xxx Created on: ddmmmyy hh:mm


Similar tables will be created for T16.1.9.5.1, T16.1.9.5.2, T16.1.9.6.1 and T16.1.9.6.2

T16.1.9.5.1 Summary of Demographic Data (Intent-to-Treat Population)

T16.1.9.5.2 Summary of Baseline Dermatological Assessment (Intent-to-Treat Population)

T16.1.9.6.1 Summary of Demographic Data (Per-Protocol Population)

T16.1.9.6.2 Summary of Baseline Dermatological Assessment (Per-Protocol Population)


Taro Pharmaceuticals U.S.A., Inc Desoximetasone Spray, 0.15% 

T16.1.9.7.1 Summary of Frequency of Investigator Global Assessment (IGA)

(Intent-to-Treat Population)

| | | Test: | Dlambor |
|---|---|---|---|
| Visit | Score | Desoximetasone<br>Topical spray, 0.15%<br>N=xx | Vehicle spray |
| | 0 (Clear) | xx (xx.x%) | xx (xx.x%) |
| | 1 (Minimal) | xx (xx.x%) | xx (xx.x%) |
| | 2 (Mild) | xx (xx.x%) | xx (xx.x%) |
| | 3 (Moderate) | xx (xx.x%) | xx (xx.x%) |
| | 4 (Severe) | xx (xx.x%) | xx (xx.x%) |
| 2 | 0 (Clear) | xx (xx.x%) | xx (xx.x%) |
| | 1 (Minimal) | xx (xx.x%) | xx(xx.x%) |
| | 2 (Mild) | xx (xx.x%) | xx(xx.x%) |
| | 3 (Moderate) | xx (xx.x%) | xx(xx.x%) |
| | 4 (Severe) | $XX (XX.X^{0/6})$ | xx (xx.x%) |
| κ4 | | | |

Path: L:\Studies\_Sas\_Codes\Clinical Trial\71542603\PDF\xxx Created on: ddmmmyy hh:mm


Novum Pharmaceutical Research Services Protocol / Study No. DSXS 1505 / 71542603 T16.1.9.7.2 Summary of Frequency of Investigator Global Assessment (IGA) Taro Pharmaceuticals U.S.A., Inc

Desoximetasone Spray, 0.15%

(Per-Protocol Population)

| 1 1 2 3 3 3 3 4 4 4 4 4 6 6 6 6 6 6 6 6 6 6 6 | 0 (Clear) 1 (Minimal) 2 (Mild) 3 (Moderate) | (%x.xx) xx<br>(%x.xx) xx | (/04 223) 223 |
|---|---|---|---|
| - 2 6 4 5 | I (Minimal)<br>2 (Mild)<br>3 (Moderate) | (0/X XX) XX | (0/Y.XX) XX |
| 1 to 4 C | 3 (Moderate) | (%x xx) xx | XX (XX.X%)<br>XX (XX.X%) |
| 4 0 | ( | xx (xx.x%) | xx (xx.x%) |
| 0 | 4 (Severe) | xx (xx.x%) | xx(xx.x%) |
| , | 0 (Clear) | xx (xx.x%) | xx (xx.x%) |
| | I (Minimal) | xx (xx.x%) | xx (xx.x%) |
| 2 | 2 (Mild) | xx (xx.x%) | xx(xx.x%) |
| m | 3 (Moderate) | xx (xx.x%) | xx (xx.x%) |
| 4 | 4 (Severe) | xx (xx.x%) | xx (xx.x%) |
| w 4 | | | |

(Proportion of Patients in each Treatment that Have Clinical Success based on IGA at Day 28±2) T16.1.9.8.1 Summary of Superiority Analysis Results of Co-Primary Efficacy Endpoint (Intent-to-Treat Population)

| | | | , | | |
|---|---|---|---|---|---|
| Treatment | Number of | Number of Patients with | Number of Number of Patients with Proportion of Patients with | Treatmen | Treatment vs. Placebo |
| Group | Patients (N) | Clinical Success (n) | Clinical Success (%) | Difference P-value | P-value |
| Placebo | XXX | XXX | %X.XX | | |
| Test | XXX | XXX | XX.X% | XX.X% | X.XXXX |

Superiority of Test over Placebo was tested at the 5% significance level (p < 0.05; using two-sided Z-test) in the ITT population using last observation carried forward (LOCF).

Path: L:\Studies\_Sas\_Codes\Clinical Trial\71542603\PDF\xxx Created on: ddmmmyy hh:mm


T16.1.9.8.2 Sensitivity Testing: Summary of Superiority Analysis Results of Co-Primary Efficacy Endpoint (Proportion of Patients in each Treatment that Have Clinical Success based on IGA at Day 28±2) (Per-Protocol Population)

T16.1.9.9.1 Summary of Frequency of Total Lesion Severity Score (TLSS)

Novum Pharmaceutical Research Services Protocol / Study No. DSXS 1505 / 71542603

(Intent-to-Treat Population)

| | | | Test: | Dlocabo |
|---|---|---|---|---|
| Signs and<br>Symptoms | Visit | Score | Desoximetasone<br>Topical spray, 0.15%<br>N=xx | Vehicle spray |
| TLSS | | 0 (Clear) | xx (xx.x%) | XX (XX.X <sup>0</sup> / <sub>0</sub> ) |
| | | 1 (Almost Clear) | xx (xx.x%) | xx (xx.x%) |
| | | 2 (Mild) | xx (xx.x%) | xx (xx.x%) |
| | | 3 (Moderate) | xx (xx.x%) | xx (xx.x%) |
| | | 4 (Severe) | xx (xx.x%) | xx (xx.x%) |
| | | 5 (Very Severe) | xx (xx.x%) | xx (xx.x%) |
| | 2 | 0 (Clear) | xx (xx.x%) | xx (xx.x%) |
| | | 1 (Minimal) | xx (xx.x%) | xx (xx.x%) |
| | | 2 (Mild) | xx (xx.x%) | xx (xx.x%) |
| | | 3 (Moderate) | xx (xx.x%) | xx (xx.x%) |
| | | 4 (Severe) | xx (xx.x%) | xx (xx.x%) |
| | | 5 (Very Severe) | xx (xx.x%) | xx (xx.x%) |
| | m | | | |
| | 4 | | | |
| Scaling | | | | |
| Erythema | | | | |
| Plaque Elevation | | | | |

Path: L:\Studies\_Sas\_Codes\Clinical Trial\71542603\PDF\xxx Created on: ddmmmyy hh:mm


T16.1.9.9.2 Summary of Frequency of Total Lesion Severity Score (TLSS) (Per-Protocol Population)

(Proportion of Patients in each Treatment that Have Treatment Success based on TLSS at Day 28±2) T16.1.9.10.1 Summary of Superiority Analysis Results of Co-Primary Efficacy Endpoint (Intent-to-Treat Population)

| Treatment | Number of | Number of Patients with | Proportion of Patients with | Treatmen | Freatment vs. Placebo |
|---|---|---|---|---|---|
| Group | Patients (N) | Patients (N) Treatment Success (n) | Treatment Success (%) | Difference P-value | P-value |
| Placebo | XXX | XXX | %X.XX | | |
| Test | XXX | XXX | %X.XX | %X:XX | x.xxxx |

Superiority of Test over Placebo was tested at the 5% significance level (p < 0.05; using two-sided Z-test) in the ITT population using last observation carried forward (LOCF).

Path: L:\Studies\_Sas\_Codes\Clinical Trial\71542603\PDF\xxx Created on: ddmmmyy hh:mm


T16.1.9.10.2 Sensitivity Testing: Summary of Superiority Analysis Results of Co-Primary Efficacy Endpoint (Proportion of Patients in each Treatment that Have Treatment Success based on TLSS at Day 28±2) (Per-Protocol Population) 

# T16.1.9.11 Summary of Percent BSA Affected by Visit

Novum Pharmaceutical Research Services Protocol / Study No. DSXS 1505 / 71542603

# (Intent-to-Treat Population)

| Visit | Statistic | Test: Desoximetasone Topical spray, 0.15% N=xx | Placebo:<br>Vehicle spray<br>N=xx |
|---|---|---|---|
| 1 (Baseline) | u | XX | XX |
| | Mean ± SD | $xxx.x \pm xx.x$ | $xxx.x \pm xx.x$ |
| | Median | xxx.x | XXX.X |
| | Range | XXX - XXX | XXX - XXX |
| 2 to 4 | | | |
| Change from Baseline to Day $28 \pm 2$ | | | |

Path: L:\Studies\_Sas\_Codes\Clinical Trial\71542603\PDF\xxx Created on: ddmmmyy hh:mm


T16.1.9.12 Summary of ANCOVA Analysis Results of Secondary Efficacy Endpoint (Change from Baseline in %BSA Affected at Day  $28\pm2$ ) (Intent-to-Treat Population)

Taro Pharmaceuticals U.S.A., Inc Desoximetasone Spray, 0.15%

| | | | | | Treatment vs. Placebo | Placebo | |
|---|---|---|---|---|---|---|---|
| Freatment | Number of | | Std Err | LSMean | Std Err | | |
| Group | Patients (N) | LSMean | LSMean | Difference | Difference | 95% CI | P-value |
| lacebo | XXX | XXX.XX | XXX.XX | | | | |
| Test | xxx | XXX.XX | XXX.XX | XXXXX | XXX.XX | XX.X - XX.X | X.XXXX |

Analysis of Covariance (ANCOVA) with treatment and site as fixed effects and baseline %BSA as a covariate in the model was used for superiority testing at the 5% significance level in the ITT population using LOCF.

Path: L:\Studies\_Sas\_Codes\Clinical Trial\71542603\PDF\xxx Created on: ddmmmyy hh:mm

### Taro Pharmaceuticals U.S.A., Inc Desoximetasone Spray, 0.15%

Novum Pharmaceutical Research Services Protocol / Study No. DSXS 1505 / 71542603

T16.1.9.13 Overall Summary of Adverse Events

| | i est: | Dle seles. | |
|---|---|---|---|
| Description | Desoximetasone<br>Topical spray, 0.15%<br>N=xx | riaceno:<br>Vehicle spray<br>N=xx | Total<br>N=xx |
| Patients Randomized | xxx | XXX | XXX |
| Patients with at least one AE | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) |
| Discontinued study drug due to above AEs | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| AEs reported | XXX | XXX | XXX |
| Mild | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) |
| Moderate | xx (xx.x%) | xx (xx.x%) | $xx (xx.x^{0})$ |
| Severe | xx (xx.x%) | xx (xx.x%) | (xx.xx) |
| Not Related | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Related | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Death | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Serious AE | xx (xx.x%) | xx (xx.x%) | (%x.xx) xx |

Path: L:\Studies\_Sas\_Codes\Clinical Trial\71542603\PDF\xxx Created on: ddmmmyy hh:mm

T16.1.9.14 Summary of Frequency of All Adverse Events by Body System

(Safety Population)

| | | Desoxi Topical s | Test: Desoximetasone Topical spray, 0.15% (N = xxx) | Plac<br>Vehicl | Placebo:<br>Vehicle spray<br>(N = xxx) | |
|---|---|---|---|---|---|---|
| Body System | MedDRA Term Events Patients | Events | Patients | Events | Events Patients | Fisher's<br>p-value |
| Patients with at least one AE Total | Total | XX | (%x.xx) xx | XX | xx (xx.x%) | X.XXXX |
| Ear and labyrinth disorders | Ear pain | × | xx (xx.x%) | × | $xx(xx.x^{0})$ | X.XXX |
| | etc. | | | | | |
| etc. | | | | | | |

Path: L:\Studies\_Sas\_Codes\Clinical Trial\71542603\PDF\xxx Created on: ddmmmyy hh:mm

# Protocol / Study No. DSXS 1505 / 71542603 T16.1.9.15 Summary of Frequency of All Adverse Events by Relationship

Taro Pharmaceuticals U.S.A., Inc Desoximetasone Spray, 0.15% (Safety Population)

Novum Pharmaceutical Research Services

| | | T<br>Desoxii<br>Topical sp<br># of) | Test: Desoximetasone `opical spray, 0.15% # of Events (N = xxx) | Plac<br>Vehicle<br># of E<br>(N = | Placebo: 'ehicle spray # of Events (N = xxx) |
|---|---|---|---|---|---|
| Body System | MedDRA Term | Related | Related Not Related | Related | Related Not Related |
| Total AEs | Total | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx(xx.x) |
| Ear and labyrinth disorders | Ear pain | XX | X | XX | XX |
| | Hypoacusis | × | XX | XX | XX |

N = Total number of events in each treatment group; Percentage is based on total number of events. Related includes "Possible", "Probable", or "Definite" related.

Path: L:\Studies\_Sas\_Codes\Clinical Trial\71542603\PDF\xxx Created on: ddmmmyy hh:mm


T16.1.9.16 Summary of Frequency of All Adverse Events by Severity

(Safety Population)

| | | D<br>Top | Test: Desoximetasone Optical spray, 0.15% # of Events (N = xxx) | ne<br>15% | ŕ | Placebo:<br>Vehicle spray<br># of Events<br>(N = xxx) | À |
|---|---|---|---|---|---|---|---|
| Body System | MedDRA Term | Mild | Moderate | Severe | Mild | Moderate | Mild Moderate Severe |
| Total AEs | Total | (%x.xx) xx | (%x.x) xx $(%x.x)$ xx $(%x.x)$ xx | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Ear and labyrinth disorders | Ear pain | XX | XX | ×× | × | ×× | × |
| | Hypoacusis | × | XX | × | XX | × | XX |

N = Total number of events in each treatment group; Percentage is based on total number of events.

Path: L:\Studies\_Sas\_Codes\Clinical Trial\71542603\PDF\xxx Created on: ddmmmyy hh:mm

T16.1.9.17 Summary of Frequency of Serious Adverse Events

### (Safety Population)

| Placebo:<br>Vehicle spray<br># Events | XX |
|---|---|
| Test: Desoximetasone Topical spray, 0.15% # Events | ×× |
| MedDRA Term | Alcohol poisoning |
| Body System | Injury, poisoning and procedural complications |

Path: L:\Studies\_Sas\_Codes\Clinical Trial\71542603\PDF\xxx Created on: ddmmmyy hh:mm

T16.1.9.18 Summary of Adverse Events by Treatment (Safety Population)

Test: Desoximetasone Topical spray, 0.15%

| | | Severity | | Relationship | Relationship to Study Drug |
|---|---|---|---|---|---|
| Body System | Mild | Moderate | Severe | Related | Not Related |
| MedDKA Lerm | n (%) | II ( ½0) | II (70) | (0/) 11 | (0/) |
| Total AEs (N=xxx) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Ear and labyrinth disorders | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Ear pain | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | $xx(xx.x^0)$ | xx (xx.x%) |
| Hypoacusis | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |

N = Total ABs in Test Group; n (%) = Number of ABs (Percent of Total ABs in Test Group) Related includes "Possible", "Probable", or "Definite" related.

Path: L:\Studies\_Sas\_Codes\Clinical Trial\71542603\PDF\xxx Created on: ddmmmyy hh:mm


Programming Note: Similar tables will be created for Placebo groups.

### Taro Pharmaceuticals U.S.A., Inc Desoximetasone Spray, 0.15%

T16.1.9.19 Summary of Vital Signs

Novum Pharmaceutical Research Services Protocol / Study No. DSXS 1505 / 71542603

| Vital Signs | Visit | Statistic | Test: Desoximetasone Topical spray, 0.15% N=xx | Placebo:<br>Vehicle spray<br>N=xx |
|---|---|---|---|---|
| Systolic Blood Pressure (mmHg) | | u | XX | XX |
| | | Mean ± SD | $XXX.X \pm XX.X$ | $xxx.x \pm xx.x$ |
| | | Median | XXXX.X | XXXX.X |
| | | Range | XXX - XXX | xxx - xxx |
| | 2 | | | |
| | m | | | |
| | 4 | | | |
| Diastolic Blood Pressure (mmHg) | | | | |
| Heart Rate (bpm) | | | | |
| Respiration Rate (rpm) | | | | |
| Temperature (F) | | | | |

Path: L:\Studies\_Sas\_Codes\Clinical Trial\71542603\PDF\xxx Created on: ddmmmyy hh:mm

### T16.1.9.20 Summary of Frequency of Application Site Reaction (Safety Population)

Novum Pharmaceutical Research Services Protocol / Study No. DSXS 1505 / 71542603

Taro Pharmaceuticals U.S.A., Inc Desoximetasone Spray, 0.15%

| Signs and<br>Symptoms | Visit | Statistic | Test: Desoximetasone Topical spray, 0.15% N=xx | Placebo:<br>Vehicle spray<br>N=xx |
|---|---|---|---|---|
| Burning | 1 | Absent<br>Mild | xxx (xx.x%)<br>xxx (xx.x%) | xxx (xx.x%)<br>xxx (xx.x%) |
| | | Moderate | (%XXX (XXXX)) XXX | xxx (xx.x%) |
| | | Severe | xxx (xx.x%) | xxx (xx.x%) |
| | 2 | | | |
| | ι. | | | |
| | 4 | | | |
| Dryness<br>Edema | | | | |
| Erosion | | | | |
| Itching<br>Pain | | | | |

Path: L:\Studies\_Sas\_Codes\Clinical Trial\71542603\PDF\xxx Created on: ddmmmyy hh:mm

L16.2.1 Listing of Discontinued Patients

Taro Pharmaceuticals U.S.A., Inc Desoximetasone Spray, 0.15%

| Treatment | Patient<br>Randomization<br>Number | Discontinuation<br>Reason | Population |
|---|---|---|---|
| Test | XXXX-XX | Withdrawal by Subject<br>Lost to Follow-up | Per-Protocol<br>Safety |

Placebo

Path: L:\Studies\_Sas\_Codes\Clinical Trial\71542603\PDF\xxx Created on: ddmmmyy hh:mm

■ Taro Pharmaceuticals U.S.A., Inc ■

Novum Pharmaceutical Research Services Protocol / Study No. DSXS 1505 / 71542603

| | 77 |
|---|---------------|
| | == |
| | _ |
| | _ |
| | v. |
| , | _ |
| Ĺ | _ |
| • | |
| - | _ |
| | o |
| | ~ |
| | × |
| | 0 |
| ٠ | |
| | 2 |
| | _ |
| ć | 7 |
| , | _ |
| ¢ | - |
| | $\overline{}$ |
| | 9 |
| | ಯ |
| | _ |
| | ing<br>Engl |
| | - |
| • | _ |
| • | 5 |
| | S |
| • | 5 |
| | S |
| | S |
| | S |
| | S |
| > | SIT 7" |
| > | SIT 7" |
| | SIT 7" |
| > | .2.2 LIS |

| Treatment<br>Group | Patient<br>Randomization<br>Number | Event Description | Population |
|---|---|---|---|
| Test | XXXX-XX | Outside Visit Window (Visit 3) Safety | Safety |
| Placebo | | | |

Path: L:\Studies\_Sas\_Codes\Clinical Trial\71542603\PDF\xxx Created on: ddmmmyy hh:mm

Taro Pharmaceuticals U.S.A., Inc Desoximetasone Spray, 0.15%

L16.2.3 Patients Excluded from the Per-Protocol Population

Novum Pharmaceutical Research Services Protocol / Study No. DSXS 1505 / 71542603

| Exclusion Reason | | Major protocol deviation |
|--------------------------|--------|--------------------------|
| Patient<br>Randomization | Number | XXXX-XX |
| Treatment | Group | Test |

Placebo

Path: L:\Studies\_Sas\_Codes\Clinical Trial\71542603\PDF\xxx Created on: ddmmmyy hh:mm

### Taro Pharmaceuticals U.S.A., Inc Desoximetasone Spray, 0.15%

| _ |
|---------------|
| Data |
| ď |
| 7 |
| .≃ |
| phic |
| g |
| 31.5 |
| ~ |
| ĕ |
| Ä |
| <u> </u> |
| بيه |
| of |
| ы |
| $\Box$ |
| := |
| . S |
| :3 |
| $\overline{}$ |
| _ |
| 4 |
| $\sim$ i |
| 2 |
| L16.2 |

Novum Pharmaceutical Research Services Protocol / Study No. DSXS 1505 / 71542603

| Treatment | Patient | | | , a | • |
|---|---|---|---|---|---|
| Crons | Randomization | Age | Gender | Ethnicity | Kace |
| dinaro | Number | | | | |
| Test | XXXX-XX | 30 | Female | Not Hispanic or Latino | Black or African American |

Placebo

Path: L:\Studies\_Sas\_Codes\Clinical Trial\71542603\PDF\xxx Created on: ddmmmyy hh:mm

## L16.2.4.2 Listing of Medical History

Taro Pharmaceuticals U.S.A., Inc Desoximetasone Spray, 0.15%

Novum Pharmaceutical Research Services Protocol / Study No. DSXS 1505 / 71542603

| T | Patient | | Diagnosis or | | | |
|---|---|---|---|---|---|---|
| reatment | Randomization | System | Surgical | Start Date | End Date | Ongoing |
| Group | Number | | Procedure | | | |
| Test | XXXX-XX | Gynecologic | Menopause | yyyy-mm-dd | yyyy-mm-dd | |

Placebo

Path: L:\Studies\_Sas\_Codes\Clinical Trial\71542603\PDF\xxx Created on: ddmmmyy hh:mm

# L16.2.4.3 Listing of Concomitant Medication

Taro Pharmaceuticals U.S.A., Inc Desoximetasone Spray, 0.15%

Novum Pharmaceutical Research Services Protocol / Study No. DSXS 1505 / 71542603

| Treatment<br>Group | Patient<br>Randomization<br>Number | Treatment<br>Area | Medication | Dosage | Frequency | Route | Start/End<br>Date | Indication |
|---|---|---|---|---|---|---|---|---|
| Test | XXXX-XX | No | Lisinopril | 20 MG QD | ΦÒ | PO | yyyy-mm-dd /<br>yyyy-mm-dd | Hypertension |

Placebo

Path: L:\Studies\_Sas\_Codes\Clinical Trial\71542603\PDF\xxx Created on: ddmmmyy hh:mm

## L16.2.5.1 Listing of Visit Date Information

Novum Pharmaceutical Research Services Protocol / Study No. DSXS 1505 / 71542603

| reatment<br>Froup | Patient<br>Randomization<br>Number | Informed<br>Consent Signed | Visit 1 | Visit 2 | Visit 3 | Visit 4 /<br>Early Termination | Visit 5<br>Follow-up |
|---|---|---|---|---|---|---|---|
| | XXXX | yyyy-mm-dd | yyyy-mm-dd | d yyyy-mm-dd | yyyy-mm-dd | yyyy-mm-dd | yyyy-mm-dd |

Placebo

Path: L:\Studies\_Sas\_Codes\Clinical Trial\71542603\PDF\xxx Created on: ddmmmyy hh:mm

# L16.2.5.2 Listing of Drug Administration

Novum Pharmaceutical Research Services Protocol / Study No. DSXS 1505 / 71542603

| Treatment<br>Group | Patient<br>Randomization<br>Number | Date of<br>First Dose | Date of<br>Last Dose | Total<br>Intended | Total<br>Doses Applied | Compliance (%) |
|---|---|---|---|---|---|---|
| Test | XXXX | yyyy-mm-dd | yyyy-mm-dd | xx | XX | XX.X |

Placebo

Note to programmer: Compliance = [Actual number of applications] / [Planned number of applications] \* 100%, where:

Planned number of applications is determined as follows:

for patients who completed the study successfully: 56 applications (28 days of twice daily dosing); for patients who discontinued early: the minimum between 56 and [(Date of Discontinuation – Date of First Application +1)\*2].

Path: L:\Studies\_Sas\_Codes\Clinical Trial\71542603\PDF\xxx Created on: ddmmmyy hh:mm

# L16.2.5.3 Listing of Study Medication Weight

Novum Pharmaceutical Research Services Protocol / Study No. DSXS 1505 / 71542603

| Treatment<br>Group | Patient<br>Randomization<br>Number | Bottle | Date<br>Dispensed | Weight<br>Dispensed<br>(g) | Date<br>Collected | Weight<br>Collected<br>(g) |
|---|---|---|---|---|---|---|
| Test | XXXX | Bottle 1 | yyyy-mm-dd | XX | yyyy-mm-dd | XX |
| | | Bottle 2 | yyyy-mm-dd | XX | yyyy-mm-dd | XX |

Placebo


Path: L:\Studies\_Sas\_Codes\Clinical Trial\71542603\PDF\xxx Created on: ddmmmyy hh:mm

L16.2.6.1 Listing of Investigator Global Assessment (IGA)

| | | | IGA* | *x | | |
|---|---|---|---|---|---|---|
| Treatment<br>Group | Patient<br>Randomization<br>Number | Visit 1 | Visit 2 | Visit 3 | Visit 4 / Early<br>Termination | Clinical<br>Success |
| Test | XXXX-XX | <i>ເ</i> ດ ເດ | m m | 7 7 | 0 71 | Success<br>Failure |

Placebo

\*IGA: 0 = Clear; 1 = Minimal; 2 = Mild; 3 = Moderate; 4 = Severe;

Path: L:\Studies\_Sas\_Codes\Clinical Trial\71542603\PDF\xxx Created on: ddmmmyy hh:mm

## Desoximetasone Spray, 0.15%

L16.2.6.2 Listing of Total Lesion Severity Score (TLSS)

Novum Pharmaceutical Research Services Protocol / Study No. DSXS 1505 / 71542603

| | | | ) | • | | | |
|---|---|---|---|---|---|---|---|
| Treatment<br>Group | Patient<br>Randomization<br>Number | Visit | Scaling* | Erythema* | Plaque<br>Elevation* | TLSS** | Treatment<br>Success |
| Test | XXXX | | 0 | 1 | 3 | 4 | |
| | | 7 | 0 | - | c | 4 | |
| | | c, | 0 | - | 3 | 4 | |
| | | 4 | 0 | | | 7 | Success |
| Placebo | | | | | | | |

\*Scaling and Erythema: 0 = Clear; 1 = Almost Clear; 2 = Mild; 3 = Moderate; 4 = Severe; 5 = Very Severe \*\* TLSS = Scaling + Erythema + Plaque elevation

Path: L:\Studies\_Sas\_Codes\Clinical Trial\71542603\PDF\xxx Created on: ddmmmyy hh:mm

Taro Pharmaceuticals U.S.A., Inc Desoximetasone Spray, 0.15%

L16.2.6.3 Listing of Psoriasis Area Severity Index (PASI), Target Lesion size and BSA Affected

| Treatment<br>Group | Patient<br>Randomization<br>Number | Visit | PASI | % BSA Affected with<br>Plaque Psoriasis | Target Lesion<br>Size<br>(cm^2) | Total<br>Baseline BSA<br>(m^2) |
|---|---|---|---|---|---|---|
| Test | × | - 0 m 4 | X X X X X | %xxx<br>%xxx<br>%xxx | XXXXX | X.XXX |

Placebo

Path: L:\Studies\_Sas\_Codes\Clinical Trial\71542603\PDF\xxx Created on: ddmmmyy hh:mm

Taro Pharmaceuticals U.S.A., Inc Desoximetasone Spray, 0.15%

L16.2.6.4 Listing of Investigator Evaluator Initials

| Treatment<br>Group | Patient<br>Randomization<br>Number | Visit | IGA | PASI | TLSS | Application Site<br>Reactions |
|---|---|---|---|---|---|---|
| Test | XXXX | 1 | ABC | XYZ | D-G | D-G |
| | | 2 | | | | |
| | | 9 | | | | |
| | | 4 | | | | |

Placebo

Path: L:\Studies\_Sas\_Codes\Clinical Trial\71542603\PDF\xxx Created on: ddmmmyy hh:mm

L16.2.7.1 Listing of Adverse Events by Treatment

| Treatment<br>Group | Patient<br>Randomization<br>Number | Body System /<br>MedDRA Term /<br>AE Term | Treatment Start/End<br>Area Date | | Severity | Relationship<br>Severity to Study<br>Drug | Outcome | Action<br>Taken | Other<br>Action (<br>Taken | SAE? |
|---|---|---|---|---|---|---|---|---|---|---|
| Test | XXXX-XX | Nervous system disorders / No<br>Headache /<br>Headache | | yyyy-mm-dd / Mild<br>yyyy-mm-dd | | Possible | Recovered Dose None No<br>Not<br>Changed | Dose<br>Not<br>Changed | None | °Z |

Placebo


Path: L:\Studies\_Sas\_Codes\Clinical Trial\71542603\PDF\xxx Created on: ddmmmyy hh:mm

Taro Pharmaceuticals U.S.A., Inc Desoximetasone Spray, 0.15%

L16.2.7.2 Listing of Application Site Reaction

| | | | | Signs | Signs and Symptoms* | ptoms* | | |
|---|---|---|---|---|---|---|---|---|
| Treatment<br>Group | Patient<br>Randomization<br>Number | Visit | Burning | Erosion | Edema | Pain | Erosion Edema Pain Itching Dryness | Dryness |
| Test | XXXX | - | 0 | 0 | 0 | | 0 | 0 |
| | | 2 | 0 | _ | 0 | 0 | 0 | 0 |
| | | E | 0 | 0 | 0 | - | 0 | 0 |
| | | 4 | 0 | 0 | 0 | _ | 0 | 7 |

Reference Placebo

\*Signs and symptoms: 0 = Absent; 1 = Mild; 2 = Moderate; 3 = Severe

Path: L:\Studies\_Sas\_Codes\Clinical Trial\71542603\PDF\xxx Created on: ddmmmyy hh:mm

L16.2.8.1 Listing of Pregnancy Test Results

| Treatment<br>Group | Patient<br>Randomization | Visit | Result |
|--------------------|--------------------------|-------|----------|
| • | Number | | • |
| Test | XXXX-XX | 1 | Negative |
| | | 4 | Negative |

Placebo

Path: L:\Studies\_Sas\_Codes\Clinical Trial\71542603\PDF\xxx Created on: ddmmmyy hh:mm

L16.2.8.2 Listing of Vital Signs

| Treatment<br>Group | Patient<br>Randomization<br>Number | Visit | Systolic BP<br>(mmHg) | Diastolic BP<br>(mmHg) | Heart Rate<br>(bpm ) | Respiration<br>Rate<br>(rpm) | Temperature<br>(F) | Height<br>(cm) | Weight<br>(kg) |
|---|---|---|---|---|---|---|---|---|---|
| Test | XXXX-XX | - | 120 | 70 | 84 | 18 | 9.86 | XXX | XXXX.X |
| | | 7 | 140 | 80 | 74 | 18 | 97.0 | | |
| | | m | | | | | | | |
| | | 4 | | | | | | | |

Placebo

Path: L:\Studies\_Sas\_Codes\Clinical Trial\71542603\PDF\xxx Created on: ddmmmyy hh:mm

### NOVUM PHARMACEUTICAL RESEARCH SERVICES STATISTICAL ANALYSIS PLAN

Desoximetasone Spray, 0.15%

Protocol / Study No. DSXS 1505 / 71542603

### 10. APPENDICES

### Appendix A: Total Body Surface Area Calculation

To calculate the Total BSA the following procedure (Mosteller Formula)<sup>21</sup> should be followed.

Total Body Surface Area (BSA) in meters squared

$$m^2 = ((height (cm) x weight (kg)) / 3600)^{1/2}$$

Patient's height and weight should preferably be measured in cm and kg however if needed:

To convert inches (in) to centimeters (cm) the following conversion should be used 1 inch = 2.54 cm

To convert pounds (lbs) to kilograms (kg) the following conversion should be used. 1 lb = 0.45 kg

The patient's height and weight should be reported to the nearest cm and nearest 0.5 kg. The BSA should be reported to the nearest second decimal place.

For example a patient who is 68 inches tall and weighs 180 lbs will have a reported BSA of:

### %BSA Affected

To calculate the %Body Surface Area Affected the "Rule of Nine" will be used.

Body Surface Area affected will be calculated using the standard medical procedure of the "Rule of Nines". The patient's palm surface of the hand represents approximately one percent of his/her body surface area. (5) Calculate to the nearest whole percentage.

### NOVUM PHARMACEUTICAL RESEARCH SERVICES STATISTICAL ANALYSIS PLAN

Desoximetasone Spray, 0.15%

Protocol / Study No. DSXS 1505 / 71542603

| Part | 10-14 year child body<br>% of total | Adult<br>body<br>% of total |
|---|---|---|
| Arm | 9.5% | 9% |
| Head | 12% | 9% |
| Neck | 1% | 1% |
| Leg | 18% | 18% |
| Anterior trunk | 16% | 18% |
| Posterior trunk | 16% | 18% |



To be eligible for inclusion in the study a patient must have a % BSA affected of 5-10%

### NOVUM PHARMACEUTICAL RESEARCH SERVICES STATISTICAL ANALYSIS PLAN

Desoximetasone Spray, 0.15%

Protocol / Study No. DSXS 1505 / 71542603

### **Appendix B: Total Lesion Severity Score (TLSS)**

| Score | Grade | Erythema | Scaling | Plaque Elevation |
|---|---|---|---|---|
| 0 | Clear | No evidence of | No evidence of | No evidence of plaques |
| | | erythema | scaling | above normal skin level |
| 1 | Almost Clear | Pink | Occassional fine | Slight, just discernable |
| | | discoloration, | scales hardly | elevation above normal |
| | | minimal erythema | noticeable | skin level |
| 2 | Mild | Light red | Slight but definite | Discernable elevation |
| | | coloration | roughness, fine scale | above normal skin level |
| | | | present, no cracking | upon examination, but |
| | | | | not pronounced |
| 3 | Moderate | Moderate redness, | Moderate roughness, | Definite plaque |
| | | but not dark | somewhat coarse | formation with |
| | | | scaling | rounded/sloped edges to |
| | | | | plaque |
| 4 | Severe | Dark red | Marked roughness, | Marked elevation with |
| | | coloration | coarse/thick scaling, | hard, distinct edges to |
| | | | cracking may be | plaque |
| | X7 C | X7 1 1 1 | evident | V |
| 5 | Very Severe | Very dark red | Very thick scales | Very marked elevation, |
| | | coloration with | covering extensive | very hard and sharp |
| | | induration present | area, severe | edges to plaque |
| | | | cracking/fissures may<br>be evident | |
| L | | | DE EVIGENT | |

To be considered for inclusion in the study, the Target Lesion must have a minimum plaque elevation score of  $\geq 2$ .

### NOVUM PHARMACEUTICAL RESEARCH SERVICES STATISTICAL ANALYSIS PLAN

Desoximetasone Spray, 0.15%

Protocol / Study No. DSXS 1505 / 71542603

### Appendix C: Investigator's Global Assessment (IGA)

To be eligible for inclusion in the study the IGA must be 2 - 3 at baseline.

| Score | Category | Description |
|---|---|---|
| 0 | Clear | Plaque: elevation: no evidence of plaque elevation above normal skin |
| | | level. |
| | | Scaling: no evidence of scaling |
| | | Erythema: no redness |
| 1 | Minimal | Plaque elevation: very slight elevation above normal skin level, easier |
| | | felt than seen |
| | | Scaling: limited amount of very fine scales partially covers some of |
| | | the plaques |
| | | Erythema: very few of the plaques are light red |
| 2 | Mild | Plaque elevation: slight but definite elevation above the normal skin |
| | | level, typically with edges that are indistinct or sloped on some of the |
| | | plaques. |
| | | Scaling: mainly fine scales, some plaques are partially covered. |
| | | Erythema: some plaques are light red |
| 3 | Moderate | Plaque elevation: moderate elevation with rounded or sloped edges on |
| | | most of the plaques |
| | | Scaling: somewhat coarser scales; most plaques are partially covered. |
| | | Erythema: most plaques are red |
| 4 | Severe | Plaque elevation: marked to very marked elevation, with hard to very |
| | | hard sharp edges on virtually all or all of the plaques. |
| | | Scaling: coarse, thick scales; virtually all or all plaques are covered; |
| | | rough surface. |
| | | Erythema: virtually all or all plaques are bright to dusky red. |

### NOVUM PHARMACEUTICAL RESEARCH SERVICES STATISTICAL ANALYSIS PLAN

Desoximetasone Spray, 0.15%

Protocol / Study No. DSXS 1505 / 71542603

### Appendix D: Psoriasis Area Severity Index (PASI)

The PASI is a composite score based on the severity of four different signs of atopic dermatitis in four different areas of the body multiplied by the percent of that specific body area affected multiplied by a weighting factor.

### Erythema, Induration, Scaling will be evaluated using the severity scale below:

0 = Clear

1 = Mild

2 = Moderate

3 = Severe

4 = Very Severe

### **PASI Score**

The PASI score is calculated as follows:

Head/neck (E + I + S) x Area x 0.1

Upper Limbs

(E + I + S) x Area x 0.2

Trunk

 $(E + I + S) \times Area \times 0.3$ 

Lower Limbs  $(E + I + S) \times Area \times 0.4$ 

PASI SCORE = SUM OF ABOVE 4 REGIONS

E: Erythema,

I: Induration

S: Scaling

Severity is based on the Investigator's assessment of individual signs and symptoms 0 = none, 1 = mild, 2 = moderate, 3 = severe, 4 = very severe using the definitions above

The % of each body region affected is scored as the variable Area above in the PASI formula. For the 4 body regions (head/neck, upper limbs, trunk and lower limbs) if the:

```
Area = 0 if % affected is 0%
```

Area = 1 if % affected is 1 to 9%

Area = 2 if % affected is 10 to 29%

Area = 3 if % affected is 30 to 49%

Area = 4 if % affected is 50 to 69%

Area = 5 if % affected is 70 to 89%

Area = 6 if % affected is 90 to 100%

PASI Score can be presented to the nearest whole number (no decimals and all numbers should be rounded, 0.5 should be rounded up to the nearest whole number). The minimum score would be 0 and the Maximum Score would be 72.

### NOVUM PHARMACEUTICAL RESEARCH SERVICES STATISTICAL ANALYSIS PLAN

Desoximetasone Spray, 0.15%

Protocol / Study No. DSXS 1505 / 71542603

### **Appendix E: Application Site Reactions**

The following application site reactions will be evaluated at each visit based on the scale provided below:

Burning Erosion Edema Pain Itching Dryness

Absent 0

Mild 1 (slight, barely perceptible)

Moderate 2 (distinct presence) Severe 3 (marked, intense)